CLINICAL TRIAL: NCT06087419
Title: A Prospective, Single-arm Clinical Study of Bridging Allogeneic Stem Cell Transplantation After Treatment With Obinutuzumab in Combination With Chidamide and Venetoclax in Relapsed/Refractory Ph-ALL and B-cell Lymphoma Patients
Brief Title: A Prospective Clinical Study of Bridging alloHSCT After Treatment With Obinutuzumab in Combination With Chidamide and Venetoclax in RR Ph-ALL and B-cell Lymphoma Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Erlie Jiang, Director, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD22-HDACi-VEN-2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; chidamide
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; venetoclax; Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- combination drug group (Experimental)
  Interventions: Drug: chidamide; Drug: Venetoclax Oral Tablet; Drug: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: chidamide — 30mg twice weekly (BIW) for induction phase (cycle1-2,28 days per cycle)
Drug: Venetoclax Oral Tablet — 400mg daily d1-14 induction phase (cycle1-2, 28 days per cycle)
Drug: Inotuzumab Ozogamicin — 0.6 mg/m2 on day 1 of cycle 1-2(28 days per cycle)

SUMMARY:
This study is a multicenter, prospective, interventional clinical trial aimed at recruiting relapsed/refractory Ph-ALL patients at multiple stem cell transplantation centers, including the Stem Cell Transplantation Center of the Chinese Academy of Medical Sciences Hematology Hospital. The anticipated enrollment is 42 subjects. The enrolled patients are planned to receive a treatment regimen of chidamide in combination with venetoclax and obinutuzumab. Patients who achieve remission will undergo allogeneic stem cell transplantation, followed by continued oral maintenance therapy with chidamide for one year post-transplantation based on the disease condition.

DETAILED DESCRIPTION:
Relapsed/refractory Ph-ALL patients who meet the inclusion criteria and provide informed consent will be enrolled in the study. They will receive combination chemotherapy with chidamide, venetoclax, and obinutuzumab. After one treatment cycle, if the patient achieves complete remission (CR) and minimal residual disease (MRD) negativity, they will proceed to the preparatory phase for allogeneic stem cell transplantation. In cases where MRD remains positive after one cycle of chemotherapy, the same regimen will be repeated for an additional cycle, followed by re-evaluation. Once MRD negativity is achieved, the patient will enter the preparatory phase for allogeneic stem cell transplantation. After successful hematopoietic recovery post-transplantation (neutrophil count >0.5×10^9/L, platelet count >50×10^9/L), chidamide 10mg qd will be added for maintenance therapy, which will be continued for one year post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of acute lymphoblastic leukemia/lymphoblastic lymphoma with negative Ph chromosome or BCR/ABL fusion gene, and surface expression of CD22 on leukemic cells. First relapse, multiple relapses, or failure to achieve hematological remission after at least 3 cycles of intensive chemotherapy.
2. Age greater than or equal to 18 years.
3. Must have adequate organ function: Renal function and liver function as follows: AST, ALT, and ALP levels less than 2 times the upper limit of normal, total bilirubin level less than 1.5 times the upper limit of normal; Creatinine clearance greater than 50 mL/min; Pancreatic function: Serum amylase not higher than 1.5 times the upper limit of normal, serum lipase not higher than 1.5 times the upper limit of normal; Normal cardiac function: Ejection fraction (EF) > 60%, pulmonary artery systolic pressure ≤ 50 mmHg.
4. HIV negative, HBV and HCV negative.
5. Eastern Cooperative Oncology Group performance status assessment (ECOG-PS) score of 0-2.
6. Informed consent must be signed before the start of the study. For participants aged 18 and above, the informed consent should be signed by the patient or their immediate family member. Considering the patient's condition, if it is not favorable for the patient to sign, the informed consent may be signed by a legal guardian or immediate family member of the patient.

Exclusion Criteria:

1. Lack of CD22 expression on the surface of leukemia cells.
2. Mixed lineage leukemia.
3. Patients with concomitant malignancies; patients assessed to have accompanying diseases that pose a severe risk to patient's life or would interfere with the completion of this study.
4. Patients with a severe (≥ Grade 3) allergy to the components and excipients of obinutuzumab, idarubicin, and venetoclax.
5. Clinically significant liver disease, such as a history of veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS); severe/uncontrolled liver disease, such as cirrhosis, decompensated liver disease, acute or chronic hepatitis.
6. Active cardiac disease, defined as any of the following: history of any cardiac or vascular disease; uncontrolled or symptomatic history of angina pectoris; myocardial infarction within 6 months prior to study entry; history of clinically significant arrhythmia requiring medication or with severe clinical symptoms; uncontrolled or symptomatic congestive heart failure (> NYHA class 2); ejection fraction below the lower limit of normal range; pulmonary artery systolic pressure > 50 mmHg on echocardiography or clinical symptoms related to pulmonary arterial hypertension.
7. Known positive serological reaction for HIV or active hepatitis C virus.
8. Presence of psychiatric disorders or other conditions that would hinder compliance with study treatment and monitoring requirements.
9. Inability or unwillingness to sign the informed consent form.
10. Pregnant or lactating females.
11. Patients deemed ineligible due to other specific circumstances as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24months
  One-year overall survival rate (OS) after allogeneic stem cell transplantation.

SECONDARY OUTCOMES:
Complete remission | 24months
  Complete remission (CR) rate following treatment with obinutuzumab in combination with chidamide and venetoclax.
relapse-free survival | 24months
  One-year relapse-free survival (RFS) after allogeneic stem cell transplantation.
Incidence of graft-versus-host disease | 24months
  Incidence of graft-versus-host disease (GVHD) following allogeneic stem cell transplantation.
Engraftment rate | 24months
  Engraftment rate post-transplantation.
Minimal residual disease rate | 24months
  Minimal residual disease (MRD) clearance rate following chemotherapy.
Bridging transplant rate. | 24months
  Bridging transplant rate.

IPD SHARING:
Plan to Share IPD: Undecided